CLINICAL TRIAL: NCT01286155
Title: Epidemiology of Barrett's Esophagus: A Population Based Study
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Principal Investigator, Prasad G. Iyer, MD, Mayo Clinic
Other Study IDs: 09-002718
Record Dates: First submitted 2011-01-26; First posted 2011-01-31 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Barrett's Esophagus; Gastroesophageal Reflux Disease (GERD); Olmsted County Resident
Keywords: Barrett's esophagus; gastroesophageal reflux disease; GERD
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- with gastroesophageal reflux disease(GERD): Subjects with gastroesophageal reflux disease (GERD)
- Non-GERD: Subjects with no history of gastroesophageal reflux disease (GERD)
- Barrett's esophagus: Subjects with confirmed barrett's esophagus in Olmsted county

SUMMARY:
To assess attitudes toward screening for esophageal adenocarcinoma (EAC) and Barrett's esophagus (BE) in the community.

To develop a population based clinical risk factor prediction model for the diagnosis of BE and identify novel risk factors for BE which would make population based screening more efficient. This will be an important first step in identifying the target population for BE screening, another crucial component of making screening feasible and efficient

ELIGIBILITY:
Inclusion Criteria:

1. Case: Olmsted county residents > 18 years old from the barrett's esophagus (BE) incidence cohort who are still alive at the time of study.
2. Control # 1 : Olmsted county residents > 18 years old that responded to a recent community based survey and reported gastroesophageal reflux (GER) symptoms at least once a week and without a known diagnosis of BE.
3. Control # 2 : Olmsted county residents > 18 years old that responded to a recent community based survey that did not report any GER symptoms and without a known diagnosis of BE.

Exclusion Criteria:

1. Cases: BE subjects who

   1. Have died prior to the start of this study;
   2. Refuse to participate;
2. Controls: respondents to the "constipation survey" who

   1. Are known to have BE;
   2. Have died prior to the start of this study;
   3. Refuse to participate; -

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Olmsted county resident
Sampling Method: Non-Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome from the survey will be the proportion of patients willing to undergo an esophageal capsule study compared to those willing to undergo an endoscopic procedure (Esophagogastroduodenoscopy or transnasal endoscopy) | 18 months

SECONDARY OUTCOMES:
Study established (age, gender, ethnicity, reflux) and potential risk factors (sleep apnea, visceral adiposity, Helicobacter pylori infection, Metabolic Syndrome)to develop a clinical risk factor model for diagnosis of Barrett's esophagus(BE). | 18 months
  Metabolic Syndrome (ATP III criteria, JAMA 2001; 285: 2486-97.) defined as a combination of clinical disorders that includes the presence of three or more of the following indicators:
  1. abdominal obesity (waist circumference > 102 cm in men, > 88 cm in women);
  2. high triglyceride level (≥ 150 mg/dL);
  3. low level of high density lipoprotein (< 40 mg/dL in men; < 50 mg/dL in women);
  4. high blood pressure (≥ 130/85 mmHg);
  5. high fasting plasma glucose (≥ 110 mg/dL).

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States